CLINICAL TRIAL: NCT00742144
Title: An Open-label Phase I Study of Ofatumumab in Japanese Patients With CD20 Positive Follicular Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: Ofatumumab in Japanese Patients With CD20 Positive Follicular Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMB111148
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Leukaemia, Lymphocytic, Chronic and Lymphoma, Follicular
Keywords: CD20 positive; Chronic lymphocytic leukemia; Follicular lymphoma; GSK1841157; Japanese patient; Ofatumumab
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — ofatumumab

ARMS (1):
- ofatumumab (Experimental): Japanese patients with CD20 positive follicular lymphoma or chronic lymphocytic leukemia
  Interventions: Drug: ofatumumab

INTERVENTIONS:
Drug: ofatumumab — Ofatumumab (GSK1841157), a clear colorless liquid, is supplied in a glass vial. Each vial contains 100mg of ofatumumab in 5mL.

SUMMARY:
This is an open-label study to evaluate safety, tolerability, efficacy and PK profile of ofatumumab monotherapy in Japanese follicular lymphoma (FL) or chronic lymphocytic leukemia (CLL) patients. subject will receive ofatumumab 8 weekly infusions.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed Informed Consent.
* Histologically confirmed relapsed or refractory CD20 positive FL grade 1-3a and 1 or more clearly demarcated lesions with a largest diameter = 1.5 cm, or CD5, CD19, CD20 and CD23 positive relapse or refractory CLL.
* Subjects must have adequate blood, liver, and kidney function.
* Subjects who passed the provided periods from the last anti-cancer treatments at screening
* ECOG Performance Status of 0-2
* Life expectancy more than 24 weeks at screening

EXCLUSION CRITERIA:

* Current and past malignancy other than FL and CLL within 5 years prior to screening.
* Known Richter's transformation
* Previous autologous stem cell transplantation within 24 weeks prior to screening
* Previous allogeneic stem cell transplantation
* Known CNS involvement
* History of significant cerebrovascular disease
* Current cardiac disease requiring medical treatment
* Chronic or ongoing active infectious disease requiring systemic treatment
* Patients with pleural effusion or ascites detectable by physical examination
* Positive serology test for any of HBsAg, anti-HBc or anti-HCV
* Known HIV positive
* Pregnant or lactating women
* Women of childbearing potential and male patients not willing to use adequate contraception

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-09-19 (Actual); Primary Completion 2009-11-18 (Actual); Study Completion 2009-11-18 (Actual)

PRIMARY OUTCOMES:
tolerability | eight weeks

SECONDARY OUTCOMES:
Adverse event,Clinical laboratory tests,Immunoglobulin,HAHA,Objective response rate,Duration of response,Progression free survival,CD5,19,20,CD23 positive cells,Complement (CH50),PK parameters, | nine months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Background] Ogura M, Hatake K, Tobinai K, Uchida T, Suzuki T, Terui Y, Yokoyama M, Maruyama D, Mori M, Jewell RC, Katsura K, Hotta T. Phase I study of ofatumumab, a human anti-CD20 antibody, in Japanese patients with relapsed or refractory chronic lymphocytic leukemia and small lymphocytic lymphoma. Jpn J Clin Oncol. 2013 May;43(5):466-75. doi: 10.1093/jjco/hyt022. Epub 2013 Feb 28. PMID 23456745
- See also: Results for study OMB111148 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/OMB111148?search=study&study_ids=OMB111148#rs